CLINICAL TRIAL: NCT05080738
Title: Investigation of Upper Extremity Home Exercises Effects on Grip Strength, Range of Motion, Activity Performance and Funcionality in Patients With Scleroderma
Brief Title: Upper Extremity Home Exercises in Patients With Scleroderma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Sebahat Yaprak Cetin,PT, Principal Investigators, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-085
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Scleroderma; System; Sclerosis
Keywords: Scleroderma; Upper extremity exercises; Home exercises; Grip strength
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Intervention Model Description: 1) Intervention Group:
  The patients in the intervention group will be asked to practice upper extremity home exercises including stretching, mobility and strengthening, as home exercises, 5 days a week for 8 weeks, which will be taught by the physiotherapist. The exercises will be performed as follows:
  1. Stretching exercises: It will be applied in the form of 10 seconds*10 repetitions for fingers, wrists, elbows and shoulders.
  2. Strengthening exercises: It will be applied as 2 sets*10 repetitions for fingers, wrists, elbows and shoulders.
  Patients will be instructed to perform the exercises according to their pain tolerance. The compliance of the patients with the exercise will be checked during this process and the evaluations will be repeated at the end of 8 weeks.
  2) Control Group: The patients in the control group will be taught the principles of joint protection and evaluations will be made again after 8 weeks.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The patients in the intervention group will be asked to practice upper extremity home exercises including stretching, mobility and strengthening, as home exercises, 5 days a week for 8 weeks, which will be taught by the physiotherapist.
  Interventions: Other: Upper Extremity Home Exercises
- Control (No Intervention): Education group:Patients will be informed about joint protection principles by a physiotherapist for once.

INTERVENTIONS:
Other: Upper Extremity Home Exercises — The exercises will be performed as follows:
  1. Stretching exercises: It will be applied in the form of 10 seconds*10 repetitions for fingers, wrists, elbows and shoulders.
  2. Strengthening exercises: It will be applied as 2 sets*10 repetitions for fingers, wrists, elbows and shoulders.
  Arms: Intervention group

SUMMARY:
Hand involvement in scleroderma leads to functional disability due to the relationship between grip strength, wrist and finger movement. The vast majority of patients report that their activities are restricted and their quality of life decreases for this reason. Literature indicate that more work is needed to continue to develop and evaluate rehabilitation interventions in this population.

This study is a randomized controlled study examining the effects of 8 weeks of upper extremity home exercises on grip strength, normal joint movement, activity performance and functionality in patients with scleroderma. In our study, it is aimed to contribute to the standardization of upper extremity exercise protocols for scleroderma patients, to increase the quality of life of patients and to increase their independence in daily living activities.

DETAILED DESCRIPTION:
The primary aim of the study is to examine the effects of upper extremity exercises on joint range of motion, grip strength, activity performance and functionality in patients with scleroderma, and thus contribute to the standardization of exercise protocols for the upper extremity in patients with scleroderma. The secondary aim of the study is to ensure the independence of scleroderma patients in their daily living activities and to increase their quality of life.

At least 46 scleroderma patients meeting the inclusion criteria will be included in the study. Demographic information form, Canadian Activity Performance Measurement (COPM), Arm, Shoulder and Hand Problems Questionnaire (DASH), Chronic Rheumatological Influence of the Hands Assessment and Measurement Score Questionnaire (SACRAH), Duruöz Hand Index (DHI) will be applied to the patients, upper extremity joint range of motion will be applied, gross and fine grip strength measurements will be made.

After the initial evaluation, patients will be randomized to intervention and control groups. Upper extremity home exercises including stretching and strengthening will be taught to the intervention group, and they will be asked to do it 5 days a week for 8 weeks. For eight weeks, the patients will be supported by the phone by the physiotherapist and it will be checked whether they do the exercises. The control group will be trained on the principles of joint protection. At the end of eight weeks, patients will have their final evaluation and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of SSc according to 2013 ACR/EULAR criteria
* Having upper extremity/hand involvement
* Voluntary and consent to participate in the study

Exclusion Criteria:

* Having a known diagnosis of additional rheumatological disease
* Diagnosis of any known non-rheumatic disease
* Existence of deformity that prevents doing the exercises
* Presence of active digital ulcer Being involved in another rehabilitation program
* Having cognitive disorder
* Failure to give consent to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Activity Performance | 8 weeks
  Canadian Activity Performance Measure (Canadian Occupational Performance Measure=COPM/COPM): COPM is a standard measurement tool used to identify an individual's activity performance problems and measure performance satisfaction. COPM is administered as a semi-structured interview. The patient is asked to identify, discuss and rank certain activities that cause him or her difficulty. The five most important issues (as chosen by the patient) are recorded and the patient is asked to indicate their perception of how well they are currently performing the task and to rate how satisfied they are with this level of performance on a scale of 1 to 10 (1-5 not able to / not at all satisfied). not staying and being able to do it very well / extremely satisfied). Performance (COPM-P) and satisfaction (COPM-S) scores are summed separately and divided by five (number of problem areas). This gives average performance and satisfaction scores.
Grip strength | 8 weeks
  Gross grip strength will be measured with a hand dynamometer (Jamar) 3 times for both hands while the patient is sitting with the elbows bent at 90 degrees near the body and the average will be taken.
  Fine grip strength will be measured and recorded with a pinchmeter as lateral, triple and fingertip.

SECONDARY OUTCOMES:
Score for Assessment and quantification of Chronic Rheumatic Affections of the Hands=SACRAH | 8 weeks
  The newly developed questionnaire SACRAH includes 23 VASs covering three symptom categories (function, joint stiffness, pain) that primarily determine the status of patients with rheumatic diseases of the hand. The first part consists of 17 questions evaluating hand function. The determined daily activities are eval
Duruöz Hand Index (Duruöz Hand Index=DHI/DEI) | 8 weeks
  It consists of 18 items evaluating hand and wrist activities. The answers are evaluated on a 6-level (0-5) Likert scale and the total score ranges from 0 to 90. The degree of difficulty of the patients in trying to perform these daily activities without using any assistive devices is scored. If the patient can perform this activity without any difficulty, it is scored 0, 1 if it can be done with little difficulty, 2 if it can be done with a little difficulty, 3 if it is very difficult, 4 if it is almost impossible to perform this activity, and 5 if it is completely impossible. The values given for each activity are summed at the end of the index and this value gives the patient's DHI value.
Range of Motion | 8 weeks
  Flexion and extension range of motion will be measured and recorded by the physiotherapist passively and actively with universal goniometer and finger goniometer at appropriate positions.
Disabilities of Arm, Shoulder and Hand questionnaire: | 8 weeks
  It consists of three parts: The first part consists of 30 questions; 21 questions assess the patient's difficulty during activities of daily living, 5 questions assess symptoms (pain, activity-related pain, tingling, stiffness, weakness), and 4 questions assess social function, work, sleep and self-confidence of the patient. In all questions, the patient marks the appropriate answer according to the 5-point Likert system (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: not at all). The scores for each section are summed and divided by the number of questions and '1' is subtracted from the result. The result found is multiplied by 25. Results from 0 to 100 are obtained from each section (0: no disability, 100: maximum disability).

CONTACTS AND LOCATIONS:
Overall Officials: Sebahat Yaprak Cetin, PhD, Principal Investigator — Akdeniz University
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study is a randomized controlled trial. Data will record on Statistical Package for the Social Sciences and the data will share wih all researches which will be included the study.

REFERENCES:
- [Result] Landim SF, Bertolo MB, Marcatto de Abreu MF, Del Rio AP, Mazon CC, Marques-Neto JF, Poole JL, de Paiva Magalhaes E. The evaluation of a home-based program for hands in patients with systemic sclerosis. J Hand Ther. 2019 Jul-Sep;32(3):313-321. doi: 10.1016/j.jht.2017.10.013. Epub 2017 Dec 1. PMID 29198478